CLINICAL TRIAL: NCT06889285
Title: Comparison of Safety and Efficacy Between Programmed Intermittent Epidural Bolus (PIEB) and Continuous Epidural Infusion (CEI) for Labour Epidural Analgesia: a Randomized Controlled Trial
Brief Title: Comparison of Safety and Efficacy Between PIEB and CEI for Labour Epidural Analgesia
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Koeh Shao Keong, Dr, Hospital Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USM/JEPeM/KK/23110826
Record Dates: First submitted 2025-03-15; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Analgesia, Epidural
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participant and clinician cant be blinded in this study in view that CADD-Solis pump used in programmed intermittent epidural bolus (PIEB) group is different from conventional infusion pump with distinct patient bolus button.
  Although participant can be blinded by introducing placebo bolus in continuous epidural infusion (CEI) group, it is unethical to do so, especially when involves obstetric patient that encounter labour pain during active phase of labor.
  Only assessor can be blinded by masking the labor epidural analgesia delivery pump (be it CADD-Solis pump or conventional infusion pump), thus to reduce bias in the observed outcome
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous Epidural Analgesia (Experimental): Epidural catheter will be connected to epidural cocktail (Bupivacaine 0.1% + Fentanyl 2mcg/ml in 50ml mixture) with the protocol as below: (directly extracted from Malaysia Pain management in Obstetrics and Gynaecology Procedure Guideline 2023)
  * Loading dose 10 ml
  * Continuous infusion: 10ml/hour
  Interventions: Procedure: Continuos epidural infusion
- Programmed Intermittent Epidural Bolus (Experimental): Patient in this group receive programmed intermittent epidural bolus (PIEB) using cocktail of Ropivacaine 0.05% + fentanyl 2mcg/ml, with 10ml cocktail loading when started, then 10ml hourly bolus, with patient controlled epidural analgesia (PCEA) - 10ml per patient request, lockout interval 10minutes.
  Interventions: Procedure: Programmed intermittent epidural bolus

INTERVENTIONS:
Procedure: Continuos epidural infusion — This group of parturient will be inserted epidural catheter at L3/L4 or L4/L5 depending on anaesthetist-in-charge justification, epidural catheter will be kept 4-5 cm in epidural space and anchored with adhesive tape. Similarly, a test dose of LA Lignocaine 2% 2ml will be given after epidural insertion. Infusion tubing will be primed in advance. Epidural catheter will be connected to epidural cocktail (Bupivacaine 0.1% + Fentanyl 2mcg/ml in 50ml mixture) with the protocol as below: (directly extracted from Malaysia Pain management in Obstetrics and Gynaecology Procedure Guideline 2023)
  * Loading dose 10 ml
  * Continuous infusion: 10ml/hour
  Arms: Continuous Epidural Analgesia
Procedure: Programmed intermittent epidural bolus — This group patient will be inserted epidural catheter at L3/L4 or L4/L5 depending on anaesthetist-in-charge justification, epidural catheter will be kept 4-5 cm in epidural space and anchored with adhesive tape. A test dose of LA Lignocaine 2% 2ml will be given after epidural insertion. CADD-Solis infusion tubing will be primed in advance. Epidural catheter will be connected to epidural cocktail (Ropivacaine 0.05% + Fentanyl 2mcg/ml in 100ml mixture) with the protocol as below:
  * Loading dose: 10ml
  * Intermittent bolus: 10ml, bolus interval 1 hour, next bolus 1 hour
  * PCEA dose: 10ml, lockout interval 10 minutes
  Arms: Programmed Intermittent Epidural Bolus

SUMMARY:
The goal of this clinical trial is to compare safety and efficacy of programmed intermittent epidural bolus (PEIB) and continuous epidural infusion (CEI) in parturients during active phase of labour.

The main questions aimed to answer are:

* Will parturient using PIEB+PCEA has lower incidence of motor block as compared to CEI during labour?
* Will parturient using PIEB + PCEA has lower local anaesthetic consumption (in mg/hr) as compared to CEI during labour?
* Will parturient using PIEB + PCEA has shorter duration of second stage labour as compared to CEI?
* Will parturient using PIEB + PCEA has better satisfaction score when compared to CEI during labour?

Participants will be randomised into PIEB group and CEI group after informed consent taken

* All participants will be taken baseline demographic data, vital signs, Bromage score, cardiotocograph prior intervention
* Labour epidural will be inserted and started on PIEB protocol or CEI protocol based on randomisation
* Participants vital signs and Bromage score will be recorded hourly till baby delivery
* In the end of delivery, total LA consumption and duration of second stage will be recorded
* Within 24 hours, participants will be interviewed on their satisfaction score on labour epidural analgesia.

Researchers will compare PIEB and CEI to see if PIEB has better safety and efficacy as compared to CEI in labour epidural analgesia.

DETAILED DESCRIPTION:
Parturient attending to labour room in Hospital Universiti Sains Malaysia and requested for labour epidural analgesia will be screened and recruited into this clinical trial. Before participation, an informed consent will be taken from parturient.

PIEB + PCEA or CEI will be used on recruited participants based on the randomised group by primary investigator. Setup of epidural cocktail infusion pump either CADD-Solis ® pump or normal infusion pump, will be done by anaesthetic officer attending the patient.

For PIEB group, ropivacaine 0.05% + fentanyl 2mcg/ml in 100ml bag will be used for epidural analgesia. For CEI group, bupivacaine 0.1% + fentanyl 2mcg.ml in 50ml will be used for epidural analgesia. Both epidural cocktails are prepared by central pharmacist in sterile technique. Participants, researcher and the anaesthetist-in-charge can't be blinded from the study in view the CADD-Solis ® pump is unique with its PCEA bolus cord.

Prior procedure, participants baseline pain score, CTG, vital signs, Bromage score will be recorded prior to epidural catheter insertion. If CTG and vital signs are reassuring, then only anaesthetist-in-charge will proceed with epidural catheter insertion.

There will be assigned two groups of patients receiving different epidural regimen;

I. PIEB + PCEA group

This group patient will be inserted epidural catheter at L3/L4 or L4/L5 depending on anaesthetist-in-charge justification, epidural catheter will be kept 4-5 cm in epidural space and anchored with adhesive tape. A test dose of LA Lignocaine 2% 2ml will be given after epidural insertion. CADD-Solis infusion tubing will be primed in advance. Epidural catheter will be connected to epidural cocktail (Ropivacaine 0.05% + Fentanyl 2mcg/ml in 100ml mixture) with the protocol as below:

* Loading dose: 10ml
* Intermittent bolus: 10ml, bolus interval 1 hour, next bolus 1 hour
* PCEA dose: 10ml, lockout interval 10 minutes

II. CEI group This group of parturient will be inserted epidural catheter at L3/L4 or L4/L5 depending on anaesthetist-in-charge justification, epidural catheter will be kept 4-5 cm in epidural space and anchored with adhesive tape. Similarly, a test dose of LA Lignocaine 2% 2ml will be given after epidural insertion. Infusion tubing will be primed in advance. Epidural catheter will be connected to epidural cocktail (Bupivacaine 0.1% + Fentanyl 2mcg/ml in 50ml mixture) with the protocol as below: (directly extracted from Malaysia Pain management in Obstetrics and Gynaecology Procedure Guideline 2023)

* Loading dose 10 ml
* Continuous infusion: 10ml/hour

During epidural catheter insertion, inadvertent spinal catheterisation or dura puncture will be reported and manged to clinician justification, meanwhile patient will be withdrawn from this study.

Participant's CTG will be recorded after epidural catheterisation. After started on epidural analgesia, participants blood pressure will be recorded every 5 mins in first 30 mins, every 15 mins for another 30 mins, then every hourly subsequently. Participants' pain score will be recorded 15 mins after epidural analgesia started, then hourly recording of pain score using Visual Analogue Scale. Similarly, Bromage score will be recorded hourly by attending labour room nurse. This monitoring follows USM epidural analgesia monitoring protocol.

Any breakthrough pain requiring physician rescue will be attended by anaesthetist-in- charge, dose and amount of local anaesthetic agent given, time of breakthrough pain will be recorded in data collection sheet. If participants have unresolved labour pain despite physician rescue bolus of drug and unable to achieve pain score of < 3, the catheter will be deemed ineffective, and the participant will be removed from the study.

Any adverse event, such as pruritus, nausea vomiting, maternal hypotension or high block will be recorded if applicable. In the end of delivery, the CADD-Solis pump/Infusion pump will be examined for total consumption of epidural cocktail in ml, its average hourly consumption, number of patient's self-administered PCEA bolus.

Obstetric and neonatal outcome, such as mode of delivery, indication for instrumental or Caesarean delivery, duration of second stage of labour and neonatal Apgar score at 1 and 5 mins will be documented in data collection sheet. The parturient will be interviewed within 24 hours of delivery by a different anaesthetist not involved in the study for overall assessment of her satisfaction with labour analgesia (graded on verbal scale from 0 = very dissatisfied to 100 = extremely satisfied)

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* ASA 2 & 3w

Exclusion Criteria:

* patient refusal
* significant comorbiddities, eg patient with heart disease, kidney diseae, neurological disoder
* contraindicated to neuraxial blockade
* allergic to local anesthetic agent or opioid
* obstetric complications, eg pre-eclampsia, leaking liqour, suspicious CTG
* morbid obesity, BMI > 40
* grandmultiparous ( > 5biths at > 20 weeks gestation)
* combined spinal epidural technique for labour epidural analgesia
* height < 145cm

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only pregnant women is eligible for this study
Enrollment: 76 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
To compare the incidence of motor block during labour between parturient with PIEB + PCEA and those with CEI. | 1 year
  Bromage score is measured hourly after epidural insertion. If there is any time when Bromage is greater than 0, then will be considered presence of motor block.

SECONDARY OUTCOMES:
To compare the duration of second stage labour between parturient with PIEB+CEA and those with CEI. | 1 year
  - From patient partogram, we will calculate duration of second stage labour for each patient (from cervical os 10cm till delivery of baby)
To compare the local anaesthetic consumption (in mg/hr) during labour between parturient with PIEB + PCEA and those with CEI | 1 year
  For PIEB+ PCEA group, the LA consumption will be retrieved from CADD-Solis pump which record total of LA use and number of patient's requested bolus. As for CEI group, its consumption can be derived from amount of LA given in the syringe and manual record where amount of physician bolus given.
To compare the satisfaction score during labour between parturient with PIEB+PCEA and those with CEI | 1 year
  Within 24 hours after delivery, parturient will be interviewed on the satisfaction score on the epidural regimen given with numerical rating scale from 0 to 100, where 0 is most unsatisfied and 100 is most satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Pakar Universiti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No